CLINICAL TRIAL: NCT03209817
Title: Effects of Tomato Supplementation on Cardiovascular Health
Brief Title: Tomato Supplementation and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Jose Lara Gallegos, Dr, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HLS-JLG-03-07-17
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red cherry tomato (Experimental): 300 grams of red cherry tomatoes per day for four weeks (each)
  Interventions: Dietary Supplement: Red cherry tomato
- Yellow cherry tomato (Experimental): 300 grams of yellow cherry tomatoes per day for four weeks (each)
  Interventions: Dietary Supplement: Yellow cherry tomato
- Control No tomato (No Intervention): No tomato products consumption

INTERVENTIONS:
Dietary Supplement: Red cherry tomato — 300 grams of cherry tomatoes per day for four weeks (each)
  Arms: Red cherry tomato
Dietary Supplement: Yellow cherry tomato — 300 grams of cherry tomatoes per day for four weeks (each)
  Arms: Yellow cherry tomato

SUMMARY:
This clinical trial aims to test the effects of consuming two types of tomato (one ordinary cherry red tomato containing lycopene, and the other a yellow cherry tomato low in lycopene), on cardiovascular risk factors including endothelial function as the primary outcome, and blood lipids, inflammatory factors and blood pressure.

In a crossover design, participants of this study will randomly consume 300g of raw cherry (red and yellow) tomatoes per day for four weeks, with a control period consuming no tomato products. Before and after each intervention, the cardiovascular outcomes mentioned above will be measured in the clinic.

DETAILED DESCRIPTION:
This study will have a randomised and crossover design of 2 interventions supplementing 300g/day of two different varieties of tomato; each of these interventions will last for 4 weeks, with a control period (no tomato consumption) of 4 weeks between these. The total study period will be 12 weeks. The target sample size for this study is 30 male participants. This study visit involve 4 study visits over a 12-week period plus a screening visit before the intervention.

In this study, the interventions will require participants to consume two different varieties of fresh tomatoes in random order. Participants will be given all the tomato to be consumed during the study, and will be instructed not to consume additional tomato sources. The amount of tomato to be consumed will be delivered every week. Participants will consume the tomatoes anytime as snack or with meal. In order to control for other dietary factors, participants will also be asked to record food diary throughout the first study period (4 weeks) and will be recommended to repeat their own dietary pattern for the control period and second study period to match up the food and nutrition intake throughout the whole study. They should not alter their usual diet and exercise patterns when completing the food diary or study. Before and after each 4 weeks intervention or control period, participant will attend the study visit for measurements.

Baseline measurements will be taken at the start of the first study period. All measurements will be measured at fasted state on before and after 4-week study period. Anthropometric measurements including height and weight, a total of 72ml venous blood samples (18ml each measurement) will be collected by researcher. Spot urine and saliva samples will be collected into a flask provided by participants themselves. Plasma and urine analyses will not commence until the full intervention study is complete, and all samples from each subject are analysed within one batch to reduce inter-batch variation. Trained researchers will obtain blood sample in this study.

Before the start of the trial, 4 volunteers will be recruited to consume 1 week of 300g red cherry tomato per day for 7 days in order to establish expected serum levels of lycopene after tomato supplementation. The aim of this is to develop cut-off serum levels to establish compliance with interventions. Six ml of fasting blood will be taken at baseline and after the 1 week consumption of red cherry tomato.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged between 18-60.
* Healthy.
* Non smoker.
* Not taking antioxidant supplement.
* No known allergy or intolerance to tomato.

Exclusion Criteria:

* Female
* Aged below 18 or above 60 years old.
* Suffering and taking medications for hypertension (>140/90mmHg), diabetes, high blood cholesterol and heart problems (e.g. arrhythmia, high-grade stenosis of the carotid artery or carotid sinus syndrome).
* Taking antioxidant supplements.
* Smoking.
* Allergy to tomato or tomato products.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation (FMD) | at 4 weeks
  To assess macrovascular endothelial function.
Laser doppler imaging (LDI) | at 4 weeks
  To assess the microvascular endothelial function.
Pulse wave velocity (PWV) and pulse wave analysis (PWA) | at 4 weeks
  To assess arterial stiffness

SECONDARY OUTCOMES:
Ambulatory blood pressure | at 4 weeks
  24 hours blood pressure
Blood lipids | at 4 weeks
  Total, LDL, HDL cholesterol and triglycerides
Interleukin-6 (IL-6) | at 4 weeks
  Interleukin-6 (IL-6)
C-reactive protein (CRP) | at 4 weeks
  C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lara, PhD, Principal Investigator — Northumbria University
Locations (1):
- Department of Applied Sciences, Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng HM, Koutsidis G, Lodge JK, Ashor A, Siervo M, Lara J. Tomato and lycopene supplementation and cardiovascular risk factors: A systematic review and meta-analysis. Atherosclerosis. 2017 Feb;257:100-108. doi: 10.1016/j.atherosclerosis.2017.01.009. Epub 2017 Jan 13. PMID 28129549